CLINICAL TRIAL: NCT00550095
Title: A 24 Week, Multi-centre, Open Label, Non Controlled Study to Assess the Efficacy of Valsartan in Reducing Albuminuria/Proteinuria in Hypertensive Patients With Type 2 Diabetes Mellitus
Brief Title: To Assess the Effects of Valsartan on Albuminuria/Proteinuria in Hypertensive Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVAL489AEG03
Record Dates: First submitted 2007-10-24; First posted 2007-10-26 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Microalbuminuria; Proteinuria
Keywords: Microalbuminuria/proteinuria; hypertensive patients with type 2 diabetes; Valsartan; microalbuminuria/proteinuria in hypertensive patients with type 2 diabetes
MeSH Terms: conditions — Proteinuria | interventions — Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): valsartan
  Interventions: Drug: valsartan

INTERVENTIONS:
Drug: valsartan

SUMMARY:
This study is designed to assess the efficacy of the different dosage forms of Valsartan[80, 160, and 320 mg] in reducing microalbuminuria/proteinuria in hypertensive patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 35 to 75.
* Type 2 diabetes mellitus (DM) patients coupled with hypertension [sitting systolic blood pressure (SSBP) 140-179 mm Hg and/or SDBP 90-109 mm Hg].
* Urinary albumin creatinine Ratio (UACR)) indicating microalbuminuria/proteinuria [30-1000 mg/g or 2.5-25 mg/mmol]
* Body mass index (BMI) <40 kg/m2
* Patients who will sign an informed consent.

Exclusion Criteria

* Type 1 DM
* All causes of secondary diabetes mellitus
* Women of childbearing potential who refuse to use contraception.
* Pregnant or lactating females.
* Severe hypertension [SSBP> 180 mmHg, sitting diastolic blood pressure (SDBP) > 110 mmHg ]
* Patients who are on combo therapy to control BP
* Patients who are already on Valsartan.
* Hypersensitivity to Valsartan.
* Renal artery stenosis [ unilateral or bilateral]
* Patients taking β blockers, (Angiotensin Converting Enzyme Inhibitor (ACEI) or spironolactone
* Heart Failure
* History of myocardial infarction, Percutaneous Transluminal Coronary Angioplasty(PTCA) or cerebrovascular accident within the preceding 3 months.
* Creatinine levels > 1.4 mg/dl [ 0.07mmol/l]. Liver enzymes > 2 times Upper Limit of the Normal Range(ULN). Diabetic keto-acidosis (DKA) within the last 6 months. Presence of diabetic neuropathy or retinopathy. Diabetic foot complications. Presence of infection at time of screening. Hyperkalemia (serum K+ > 5.5 mmol/L)

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 509 (Actual)
Dates: Start 2007-06; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Change in Albumin Creatinine Ratio (ACR) from baseline over a period of 24 weeks. | Week 24

SECONDARY OUTCOMES:
Percent reduction of (BP) at 24 weeks compared to baseline level. Percent of patients whose BP is controlled at 24 weeks (< 130/80) | Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Sponsor GmbH
Locations (1):
- Novartis Investigative Site ,, Cairo, Egypt